CLINICAL TRIAL: NCT04324476
Title: A Multicenter Phase II Clinical Study of Bevacizumab Combined With Biweekly XELOX/XELIRI Alternative First-line Treatment for Unresectable Advanced Colorectal Cancer
Brief Title: A Study of Bevacizumab Plus XELOX/XELIRI for First-line Treatment in Unresectable Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Liangjun Zhu M.M., Ward Director of Internal Medicine, Jiangsu Cancer Institute & Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS-GI1902
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Advanced Colorectal Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alternating Bevacizumab plus XELOX and Bevacizumab plus XELIRI (Experimental): Induction chemotherapy:
  Alternating Bevacizumab plus XELOX and Bevacizumab plus XELIRI:
  Bevacizumab: 5mg/kg, iv, 30min, d1, 2w; Oxaliplatin: 85mg/㎡, iv, 120min, d1, 4w; Irinotecan: 150mg/㎡, iv, 90min, d15, 4w; Capecitabine: 1000mg/㎡, bid, d2-8, 2w.
  Maintenance chemotherapy:
  Bevacizumab: 7.5mg/kg, iv, 30min, d1, q3w; Capecitabine: 1000mg/㎡, bid, d2-15, 2w.
  Interventions: Drug: Bevacizumab、Oxaliplatin、Irinotecan、Capecitabine

INTERVENTIONS:
Drug: Bevacizumab、Oxaliplatin、Irinotecan、Capecitabine — Drug: Bevacizumab 5mg/kg, iv, 30min, d1, 2w; Drug: Oxaliplatin 85mg/㎡, iv, 120min, d1, 4W; Drug: Irinotecan 150mg/㎡, iv, 90min, d15, 4w; Drug: Capecitabine 1000mg/㎡, bid, d2-8, 2w.

SUMMARY:
The objective is to investigate the efficacy and safety of two-weekly alternative regimen of Bevacizumab plus XELOX/XELIRI for First-line Treatment in Unresectable Advanced Colorectal Cancer.

DETAILED DESCRIPTION:
XELOX is a commonly used chemotherapy regimen, and XELIRI has also been widely used in the second-line treatment. XELOX and XELIRI adopt the three-week regimen, and the single dose of oxaliplatin and irinotecan is large, which has a great impact on the gastrointestinal toxicity and blood toxicity of patients. Therefore, there is no lack of a two-week improved regimen with increased frequency and reduced single dose applied in clinical, so that it has good safety, exact efficacy and increase the drug delivery density. Based on the above, we should not only consider the efficiency of the three drugs, but also control the toxic reaction. The objective is to evaluate the efficacy and safety of two-weekly alternative regimen of Bevacizumab plus XELOX/XELIRI for First-line Treatment in Unresectable Advanced Colorectal Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old;
2. Patients with advanced colorectal adenocarcinoma diagnosed by histopathology, or with metastasis more than 12 months after radical operation, and the metastasis could not be removed;
3. ECOG score ≤ 2, estimated survival time ≥ 3 months;
4. Leucocytes ≥ 3.5 × 109 / L, neutrophils ≥ 1.5 × 109 / L, hemoglobin ≥ 100g / L, platelets ≥ 80 × 109 / L, serum liver enzyme in patients without liver metastasis is not higher than 2.5 times of the upper limit of normal value, serum liver enzyme in patients with liver metastasis is not higher than 5 times of the upper limit of normal value, serum bilirubin level is not higher than 1.5 times of the upper limit of normal value, serum creatinine level is not higher than 1.5 times of the upper limit of normal value;
5. At least one lesion can be measured by CT or MRI;
6. No other history of malignant tumor;
7. Those who are fertile but willing to take contraceptive measures;
8. Sign the written informed consent.

Exclusion Criteria:

1. Patients with allergic, hypersensitive constitution and autoimmune diseases;
2. There are only unmeasurable lesions, such as hydrothorax and ascites, carcinomatous lymphangitis, diffuse liver invasion and bone metastasis; No measurable or non assessable lesions;
3. Pregnant or lactated women;
4. Uncontrolled symptomatic brain metastasis or mental disorder can not correctly describe subjective symptoms;
5. Major organ failure;
6. Affecting drug administration, absorption, distribution, metabolism, excretion, etc. the patient has uncontrollable epileptic attack, central nervous system disorder or loss of self-knowledge due to mental disease, physiological or pathological malnutrition, chronic diarrhea, and cachexia;
7. Patients with complete or incomplete ileus；
8. Patients with serious heart disease or history, including documented history of congestive heart failure, high-risk uncontrolled heart rate disorder, angina requiring drug treatment, clinically clear history of heart valve disease, serious myocardial infarction and stubborn hypertension;
9. Severe uncontrollable infection;
10. Alcohol and /or drug abuse or poor compliance of the investigator's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival 1 (PFS 1) | 28 months

SECONDARY OUTCOMES:
Progression Free Survival 2 (PFS 2) | 28 months
Objective Response Rate (ORR) | 28 months
Overall Survival (OS) | 28 months
The occurrence of adverse reactions (AEs) | 28 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Liangjun, Study Chair — Jiangsu Cancer Institute & Hospital
Locations (1):
- Jiangsu Cancer Institute & Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Li S, Li X, Xu H, Huang J, Zhu J, Peng Y, Bao J, Zhu L. Alternating modified CAPOX/CAPIRI plus bevacizumab in untreated unresectable metastatic colorectal cancer: a phase 2 trial. Signal Transduct Target Ther. 2024 Dec 11;9(1):346. doi: 10.1038/s41392-024-02048-z. PMID 39658608